CLINICAL TRIAL: NCT05794529
Title: Characterizing Tissue Protein Synthesis Rates of Non-small Cell Lung Carcinomas in Lung Cancer Patients
Brief Title: Lung Tumor Protein Synthesis Rates in Lung Cancer Patients
Acronym: LungMaas
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METCZ20220060
Record Dates: First submitted 2023-03-15; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patient: Lung cancer patients diagnosed a non-small cell lung carcinoma requiring resection surgery.
  Interventions: Other: There are no interventions in the present study

INTERVENTIONS:
Other: There are no interventions in the present study — There are no interventions in the present study

SUMMARY:
The current study will recruit lung cancer patients to measure tissue protein synthesis rates of non-small cell lung carcinomas and healthy lung tissue. The protein synthesis rates of healthy lung tissue will be compared to lung tumor tissue to establish the remodeling characteristics of healthy versus cancerous lung tissues. We will also examine whether tissue protein synthesis rates of non-small cell lung carcinomas are associated with various tumor- (i.e., size, subclassification) and patient-derived (i.e., inflammation, lung function, smoking status, and smoking history) parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Compos mentis
3. Diagnosed with lung cancer, with treatment requiring a thoracotomy or VATS lobectomy

Exclusion Criteria:

1. Neoadjuvant chemo- or radiotherapy in the past four weeks
2. Use of systemic steroids in the past four week
3. Insulin-dependent diabetes mellitus
4. Pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In total, we will recruit 30 lung cancer patients (diagnosed with a NSCLC) scheduled to undergo surgery. The nature and the risks of the experimental procedures will be explained to all subjects before their informed consent will be obtained. All subjects will be recruited through contact with their Surgeon at the Department of surgery at Zuyderland Medical Centre, Heerlen.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Lung tumor fractional synthetic rate | 5 days prior to surgery
  units: % per day
Lung tissue fractional synthetic rate | 5 days prior to surgery
  units: % per day
Muscle tissue fractional synthetic rate | 5 days prior to surgery
  units: % per day

SECONDARY OUTCOMES:
Plasma glucose concentrations | Baseline
  units: mmol/L
Plasma insulin concentrations | Baseline
  units: pmol/L
Plasma GH concentrations | Baseline
  units: mU/L
Plasma IGF-1 concentrations | Baseline
  units: nmol/L
Plasma IGFBP-1 concentrations | Baseline
  units: ug/L
Plasma IGFBP-3 concentrations | Baseline
  units: ug/L
Plasma CRP concentrations | Baseline
  units: mg/L
Plasma IL-1 concentrations | Baseline
  units: ng/L
Plasma IL-6 concentrations | Baseline
  units: ng/L
Plasma IL-10 concentrations | Baseline
  units: ng/L
Plasma TNF-alpha concentrations | Baseline
  units: ng/L

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share data with other researchers.